CLINICAL TRIAL: NCT06855940
Title: Evaluation of the Tooth Sensitivity and Whitening Effects of Calcium, Hydroxyapatite and Fluoride Containing Tooth Whitening Agents
Brief Title: Evaluation of Tooth Sensitivity and Whitening Effects of Different Content Teeth Whitening Agents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Tokat (Other)
Collaborators: TC Erciyes University (Other); Scientific Research Projects (Unknown)
Responsible Party: Sponsor-Investigator, Betül Tokat, research assistant, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EU-DHF-BT-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers; Discoloration of Teeth; Bleaching Sensitivity
Keywords: Bleaching Agents; Bleaching agent ( BOOST 40%); Bleaching teeth; Discoloration of Teeth; Sensitivity, Tooth
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity | interventions — Bleaching Agents

STUDY DESIGN:
Intervention Model Description: Group A: X bleaching agents Group B: Y bleaching agents Group C: Z bleaching agents
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (Active Comparator): 20 random patients( Whitening agent containing fluoride and 40% active ingredients)
  Interventions: Other: Bleaching Agents
- Group B (Active Comparator): 20 random patients(Whitening agent containing calcium and 35% active ingredients)
  Interventions: Other: Bleaching Agents
- Group C (Active Comparator): 20 random patients(Whitening agent containing hydroxyapatite and 18% active ingredients)
  Interventions: Other: Bleaching Agents

INTERVENTIONS:
Other: Bleaching Agents — whitening agent containing fluoride and 40% hydrogen peroxide
  Arms: Group A
Other: Bleaching Agents — whitening agent containing calcium and 35% hydrogen peroxide
  Arms: Group B
Other: Bleaching Agents — whitening agent containing hydroxyapatite and 18% hydrogen peroxide
  Arms: Group C

SUMMARY:
The goal of this clinical study is to evaluate the success of different whitening agents in whitening teeth in healthy volunteers aged 18-50. Also, patients' tooth sensitivity will be assessed after application. The main questions it aims to answer are:

Is the teeth whitening success of different whitening agents similar? Did participants develop tooth sensitivity to whitening agents? The researchers will compare the whitening success of 3 different whitening agents and changes in tooth sensitivity within 1 year after application.

Participants:

Whitening agent will be applied in the clinic Visit our clinic for checkups and records after 1 week, 2 weeks, 1 month, 2 months, 4 months , 6 months and 1 year after application

DETAILED DESCRIPTION:
The participants in the study were healthy volunteers between the ages of 18-50. The number of volunteers was determined by using other studies similar to this study. There are 60 volunteers in three groups, 20 volunteers in each group. A different whitening agent is applied to each group by the researcher.

The researcher did not include volunteers with poor oral hygiene, smoking, tooth sensitivity, caries, or medication use in the study.

The researcher began the study by performing color measurement and sensitivity assessment before the procedure. Then he applied the whitening agent. The volunteers who underwent the whitening procedure will be evaluated in terms of both color measurements and sensitivity changes at the end of the treatment, 1st week, 2nd week, 1st month, 2nd month, 4th month, 6th month, and 1st year control sessions.

Each patient has their own evaluation form. There are different fields for both color and sensitivity in the form according to the control dates. All numerical data are recorded in their own fields.

ELIGIBILITY:
Inclusion Criteria:

* Vital teeth
* Healthy gums
* No tooth sensitivity
* External discoloration ( tea,coffee..)
* Good oral hygiene
* No allergy to the material to be used

Exclusion Criteria:

* Decayed and devital teeth
* Presence of gingival bleeding
* History of trauma
* Presence of fractures, cracks and aesthetic restoration
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2025-10-13 (Estimated)

PRIMARY OUTCOMES:
Change in tooth color within 1 year after whitening | through study completion, an average of 1 year
  Measurement and recording of numerical values of tooth color with vita easyshade device
Change in tooth sensitivity after whitening within 1 year | through study completion, an average of 1 year
  Numerical measurement of sensitivity after bleaching with VAS (visual analog scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The work is not yet complete

REFERENCES:
- [Result] Matis BA. Tray whitening: what the evidence shows. Compend Contin Educ Dent. 2003 Apr;24(4A):354-62. PMID 12793212
- [Result] Meireles SS, Heckmann SS, Santos IS, Della Bona A, Demarco FF. A double blind randomized clinical trial of at-home tooth bleaching using two carbamide peroxide concentrations: 6-month follow-up. J Dent. 2008 Nov;36(11):878-84. doi: 10.1016/j.jdent.2008.07.002. Epub 2008 Aug 22. PMID 18722039
- [Result] Auschill TM, Hellwig E, Schmidale S, Sculean A, Arweiler NB. Efficacy, side-effects and patients' acceptance of different bleaching techniques (OTC, in-office, at-home). Oper Dent. 2005 Mar-Apr;30(2):156-63. PMID 15853099